CLINICAL TRIAL: NCT03111069
Title: A Phase I Study of Doxorubicin and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) and Intraoperative Brachytherapy for Unresectable or Refractory Pelvic and Abdominal Rhabdomyosarcoma and Undifferentiated Sarcomas in Children
Brief Title: Study of Doxorubicin and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) and Intraoperative Brachytherapy for Unresectable or Refractory Pelvic and Abdominal Rhabdomyosarcoma and Undifferentiated Sarcomas in Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI withdrew study
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0756; NCI-2018-01216 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Malignant Neoplasms of Mesothelial and Soft Tissue; Rhabdomyosarcoma, Pelvic; Rhabdomyosarcoma, Abdominal
Keywords: Malignant neoplasms of mesothelial and soft tissue; Pelvic and Abdominal Rhabdomyosarcoma; Undifferentiated Sarcomas; Unresectable or Refractory; Abdominal tumors; Hyperthermic intra-peritoneal chemotherapy; HIPEC; Abdominal surgery; Doxorubicin; Doxorubicin Hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex; Intra-operative radiation; IORT; Brachytherapy
MeSH Terms: conditions — Rhabdomyosarcoma; Abdominal Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resectable Intra-Abdominal/Pelvic Tumors (Experimental): Participants receive complete surgical tumor resection with no gross residual disease, followed by hyperthermic intra-peritoneal chemotherapy (HIPEC) using Doxorubicin.
  Interventions: Procedure: Abdominal Surgery; Drug: Doxorubicin
- Unresectable Intra-Abdominal/Pelvic Tumors (Experimental): Participants receive debulking surgery followed by intra-operative radiation (IORT) in the form of brachytherapy to the gross residual pelvic tumor sites.
  Participants have the option of returning for HIPEC 4 weeks (or more) after IORT, if active disease remains.
  Interventions: Procedure: Abdominal Surgery; Radiation: Intra-Operative Radiation

INTERVENTIONS:
Procedure: Abdominal Surgery — Resectable Intra-Abdominal/Pelvic Tumors Group: Participants receive peritonectomy, omentectomy, cytoreduction, (complete surgical tumor resection, no gross residual disease).
  Unresectable Intra-Abdominal/Pelvic Tumors Group: Participants receive debulking surgery (90% resection) , with no more than 5mm thick residual implants, totaling no more than 2.5cm2 of residual tumor.
Drug: Doxorubicin — Dose Escalation: Heated Doxorubicin delivered by Hyperthermic Intraperitoneal Chemotherapy (HIPEC). After abdominal surgery two large bore catheters are placed in the peritoneal cavity through the incision. Starting dose of Doxorubicin is 15 mg/L of HIPEC perfusate.
  Dose Expansion Starting Dose: MTD from Dose Escalation.
  Other Names: Doxorubicin Hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex
  Arms: Resectable Intra-Abdominal/Pelvic Tumors
Radiation: Intra-Operative Radiation — Standard dose brachytherapy delivered to the residual pelvic tumor sites.
  Other Names: IORT
  Arms: Unresectable Intra-Abdominal/Pelvic Tumors

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of heated doxorubicin that can be given to patients during surgery with abdominal tumors. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Surgery and Study Drug Administration:

If participant is found to be eligible to take part in this study, surgery will be performed to try to remove as many tumors from participant's abdomen as possible. The surgery is not being performed specifically for this research study and would be performed as part of participant's standard of care treatment even if participant didn't take part in this study. Participant will be given a separate consent form to sign that explains the details and risks of the abdominal surgery in more detail.

During the surgery, if it is decided that all of the tumors can be removed, the abdomen will be closed with a plastic tube left in place. Then, the abdominal wash will begin. During the wash, a pump that is connected to the plastic tube pushes the heated doxorubicin into the abdomen and then pulls it out to recirculate the doxorubicin. The heated doxorubicin will be recirculated in and out of the abdomen over 90 minutes while the surgeon gently presses on the abdomen to help the doxorubicin reach all areas in the abdomen. The plastic tube that the heated doxorubicin will be pumped through will stay in place after the surgery to drain the extra fluid. These are the same plastic tubes that would be present even if participant did not agree to take part in this study.

There is a chance that the surgeon may decide during the surgery that the abdominal wash will not be performed, for example if the disease has spread to or attached to certain organs. If this occurs, as many of the tumors will be removed as possible, followed by brachytherapy and the implantation of radioactive seeds. To perform brachytherapy, straws loaded with radioactive seeds will be inserted into the abdominal area. The radiation will then take place in the operating room over about 20 minutes. The straws will be removed before ending the surgery. Participant may be able to return for the abdominal wash procedure 4 weeks after the seeds have been implanted.

Pharmacokinetic Testing:

During participant's surgery, extra blood (about ½ teaspoon each time) and fluid from the abdominal area will be collected for pharmacokinetic (PK) testing when participant begins to receive the first infusion of the heated doxorubicin then 30, 60 and 90 minutes after the infusion has started, and again 24 hours after receiving the heated doxorubicin. The blood and fluid from the abdominal area will be collected through already placed catheters, so no additional needle sticks will be required. PK testing measures the amount of study drug in the body at different time points.

Length of Study:

Participant will remain on study for up to 6 months. Participant will be taken off study if the disease gets worse.

If the study doctor learns that the disease has come back or gotten worse at the 6 month follow-up visit, participant may be eligible to have the operation with heated doxorubicin wash repeated. If participant is eligible to have the surgery repeated, participant's active participation on this study will end and then participant will be given a new consent form to sign in order to be re-enrolled back onto this study.

Study Visits:

On Days 1-5, 11, and 14, (Day 1 being the day after surgery):

* Blood (about 1 teaspoon) will be drawn for routine tests.
* Participant will have a physical exam.

Follow-Up Visits:

About 1, 3, and 6 months after the surgery is complete, participant will have a follow-up visit and the following tests and procedures will be performed:

* Participant will have a physical exam.
* Blood (about 1-3 teaspoons) will be drawn for routine tests.
* Participant will have an ECHO to check your heart function.

It is recommended that participant has follow-up visits at MD Anderson at 3 and 6 months after surgery. In addition to blood draws (about 1-3 teaspoons each time), participant will have an MRI, CT, or PET-CT scan to check the status of the disease. These 3 and 6 month visits after surgery may be performed at participant's local doctor's office and/or laboratory.

This is an investigational study. Doxorubicin is FDA-approved and commercially available. The use of a heated doxorubicin wash during abdominal surgery in patients with tumors is investigational. The study doctor can explain how the study drug is designed to work.

Up to 28 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-6 years inclusive
2. Histologically proven RMS (with fusion status) or undifferentiated sarcoma of the pelvis or abdomen, group 3 (as defined by the IRS, intergroup rhabdomyosarcoma study group staging system seen in addendum 1)
3. Radiologic workup must demonstrate that the disease is confined to the abdominal cavity and/or is not metabolically active on PET (Positron Emission Tomography scan), outside of the abdominal cavity.
4. Patients must have a minimum expected duration of survival of greater than 6 weeks as determined and documented by the attending surgeon or medical oncologist.
5. Patients must not have any systemic illness which precludes them from being an operative candidate as determined by anesthesia preoperative evaluation. This includes but is not limited to, sepsis, liver failure, renal failure, cardiovascular failure, pulmonary failure.
6. Patients must have fully intact mental status and normal neurologic abilities. Intact mental status is defined by 'the capacity to identify and recall one's identity and place in time and space. Assessment of mental status and documentation of fully intact mental status by pediatric criteria, will be completed using physical and mental exam by the referring doctor or oncologist.
7. Patients must have adequate renal function defined as creatinine clearance or radioisotope GFR (glomerular filtration rate) >/=70mL/min/1.73m^2 or a serum creatinine based on age/gender less than the listed value in the table below: 1 to <2 years 0.6mg/dL for both males and females, 2 to <6 years 0.8mg/dL for both males and females, 6 to <10 years 1.0mg/dL for both males and females
8. Patients will be eligible if the WBC (white blood cell count) is ≥2000/µl or ANC (absolute neutrophil count) is ≥1,500 and platelets are ≥ 100,000/mm3
9. Patients will be eligible if serum total bilirubin and liver enzymes are ≤ 2 times the upper limit of normal
10. Patients must be recovered from any toxicity from all prior chemotherapy, immunotherapy, or radiotherapy and be at least 14 days past the date of their last treatment

Exclusion Criteria:

1. Patients will be ineligible if they have any concomitant cardiopulmonary disease which would place them at unacceptable risk for a major surgical procedure
2. Patients will be ineligible if they have disease outside of the abdominal cavity which is uncontrolled or PET avid.
3. Patients will be ineligible if they have a baseline neurologic toxicity of Grade 3 or greater.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Doxorubicin and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) | 1 day
  MTD defined as the highest dose in which 1 or fewer patients in 6 treated experience a dose limiting toxicity (DLT).
  Hematologic DLT defined as Grade IV neutropenia, anemia, or thrombocytopenia per Common Toxicity Criteria. Non-hematologic DLT is any Grade III or IV non-hematologic toxicity excluding Grade III nausea or vomiting, Grade III hepatic toxicity which returns to Grade I within two weeks of the HIPEC, or before hospital discharge, or Grade III fever occurring after the HIPEC per Common Toxicity Criteria.

SECONDARY OUTCOMES:
Progression of Disease | 6 months
  Disease progression defined by radio graphically visible nodules greater than 1.5 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hayes-Jordan, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org